CLINICAL TRIAL: NCT05103462
Title: Observational Study of Telehealth Physical Therapy Provided for Persons With Chronic Low Back Pain
Brief Title: Telehealth Physical Therapy for Chronic Back Pain - Ancillary Study to NCT03859713
Acronym: TeleOPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Julie Fritz, Distinguished Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00116150
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain
Keywords: Telehealth; Physical therapy; Chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal cohort design
Masking Description: The study has only one arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Physical Therapy (Experimental): Weekly sessions of education, advice and exercise instruction provided by a licensed physical therapist using real-time, interactive video conferencing platform.
  Interventions: Behavioral: Telehealth Physical Therapy

INTERVENTIONS:
Behavioral: Telehealth Physical Therapy — Weekly sessions of physical therapy provided using two-way, interactive, video technology consisting of education, advice and exercise instruction.

SUMMARY:
This study evaluated the feasibility of an 8-week physical therapy program for persons with chronic low back pain provided entirely using telehealth with real-time, interactive video sessions with a physical therapist.

DETAILED DESCRIPTION:
At the time of the onset of the COVID pandemic, the research team was conducting a clinical trial (the OPTIMIZE trial) investigating different nonpharmacologic treatments for persons with chronic low back pain (NCT03859713). One intervention arm in this trial is in-person physical therapy. COVID-related restrictions on in-person care prompted suspension of the OPTIMIZE trial. In order to accommodate persons in the midst of receiving treatment at the time of suspension, the study team adapted the in-person protocol for physical therapy for telehealth delivery using two-way, real-time video sessions. Because of the lack of research examining the feasibility of telehealth physical therapy provided in this manner, the study team decided to conduct a pilot study to examine the feasibility of the telehealth protocol.

This study was a prospective, longitudinal cohort of persons with chronic LBP seeking care in one of three healthcare systems; University of Utah Health and Intermountain Healthcare in Salt Lake City, Utah, and Johns Hopkins Medicine in Baltimore, Maryland. All participants were offered up to 8 weekly sessions of telehealth physical therapy. Outcomes included measures of acceptability, appropriateness, feasibility and fidelity as well as effectiveness measures including the Oswestry Disability Index and the PROMIS-29 health domains. Assessments occurred at baseline and after 10- and 26-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 64 years at the time of enrollment.
* Meets NIH Task Force definition of chronic LBP based on two questions: 1) How long has LBP has been an ongoing problem for you? and 2) How often has LBP been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1, and "at least half the days in the past 6 months" to question 2 is required to satisfy the NIH definition of chronic LBP.
* Healthcare visit for LBP in the past 90 days.
* At least moderate levels of pain and disability requiring ODI score >24 and pain intensity rating > 4.

Exclusion Criteria:

* Evidence of serious pathology as a cause of LBP including neoplasm, inflammatory disease (e.g., ankylosing spondylitis), vertebral osteomyelitis, etc.
* Evidence of a specific spinal pathology as the cause of LBP including spine fracture, spinal stenosis, radiculopathy, etc.
* Knowingly pregnant
* Unable to participate in telehealth due to lack of technology or internet access
* Has received physical therapy for LBP in prior 90 days
* Currently receiving substance use disorder treatment
* Any lumbar spine surgery in the past year.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Participant Satisfaction with Telehealth Treatment | 10-weeks
  Survey of participants evaluating treatment satisfaction
Rate of refusal to participate | Baseline
  Ratio of persons entering the study among all those eligibility for enrollment
Rate of enrolled participants initiating telehealth treatment | 10-weeks
  Ratio of persons attending at least 1 treatment session among all those enrolled
Number of sessions | 10-weeks
  Number of telehealth physical therapy sessions attended
Change in Oswestry from baseline to 10-weeks | baseline, 10 weeks
  10 item measure of back pain-related disability
Change in Oswestry from baseline to 26-weeks | baseline, 26 weeks
  10 item measure of back pain-related disability
Change in Pain Interference from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Pain Interference from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Pain Intensity from baseline to 10 weeks | baseline, 10 weeks
  PROMIS single item (part of PROMIS-29) assessing pain intensity on 0-10 rating scale
Change in Pain Intensity from baseline to 26 weeks | baseline, 26 weeks
  PROMIS single item (part of PROMIS-29) assessing pain intensity on 0-10 rating scale
Change in Fatigue from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Fatigue from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Sleep Disturbance from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Sleep Disturbance from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Anxiety from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Anxiety from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Depression from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Depression from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Social Role Participation from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Social Role Participation from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Physical Function from baseline to 10 weeks | baseline, 10 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Physical Function from baseline to 26 weeks | baseline, 26 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Change in Pain Self-Efficacy Scale from baseline to 10 weeks | baseline, 10 weeks
  10-item measure of confidence in performing activities even with pain
Change in Pain Self-Efficacy Scale from baseline to 26 weeks | baseline, 26 weeks
  10-item measure of confidence in performing activities even with pain

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fritz, PT, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Intermountain Health Care, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skolasky RL, Wegener ST, Aaron RV, Ephraim P, Brennan G, Greene T, Lane E, Minick K, Hanley AW, Garland EL, Fritz JM. The OPTIMIZE study: protocol of a pragmatic sequential multiple assessment randomized trial of nonpharmacologic treatment for chronic, nonspecific low back pain. BMC Musculoskelet Disord. 2020 May 11;21(1):293. doi: 10.1186/s12891-020-03324-z. PMID 32393216
- [Derived] Fritz JM, Minick KI, Brennan GP, McGee T, Lane E, Skolasky RL, Thackeray A, Bardsley T, Wegener ST, Hunter SJ. Outcomes of Telehealth Physical Therapy Provided Using Real-Time, Videoconferencing for Patients With Chronic Low Back Pain: A Longitudinal Observational Study. Arch Phys Med Rehabil. 2022 Oct;103(10):1924-1934. doi: 10.1016/j.apmr.2022.04.016. Epub 2022 Jun 3. PMID 35667399